CLINICAL TRIAL: NCT00728624
Title: Expert Group On Antibiotic Susceptibility Testing [EGAST] 2008: A Non-Interventional, Multicenter In-Vitro Study To Evaluate The Prevalence Of Beta-Lactamase Producing Strains Among Clinical Isolates Obtained From Hospital In-Patients And Comparison Of Antimicrobial Susceptibility Using Disc-Diffusion Method
Brief Title: Assessing Prevalence Of Beta Lactamase Production From Clinical Isolates Of Hospitalized Patients And Comparison Of Antibiotic Susceptibility Patterns
Acronym: EGAST 2008
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A1891005
Record Dates: First submitted 2008-08-04; First posted 2008-08-06 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Infection
Keywords: Antibiotic susceptibility; beta lactamase; ESBLs
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
EGAST 2008 is a prospective, non interventional, multicentric study (approximately 2000 isolates from 15- 20 sites).

Objectives:

* Comparison of antimicrobial susceptibility using disc-diffusion method
* Assessing prevalence of beta-lactamase producing strains among clinical isolates obtained from hospital in-patients

DETAILED DESCRIPTION:
n/a n/a

ELIGIBILITY:
Inclusion Criteria:

Isolates (as specified in the observational plan) from hospitalised patients

Exclusion Criteria:

Isolates obtained from outpatients will not be included for the study. Isolates from repeat cultures performed during in-patient follow-up that were previously recruited into the study will be excluded.

Isolates identified as commensals or contaminants will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Isolates from hospitalised patients
Sampling Method: Non-Probability Sample
Enrollment: 2039 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Comparison of antimicrobial susceptibility using disc-diffusion method | duration of trial

SECONDARY OUTCOMES:
Assessing prevalence of beta-lactamase producing strains among clinical isolates obtained from hospital in-patients | duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- India (9):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Manipal, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Chandigarh, Punjab
  - Pfizer Investigational Site, Porur, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Kolkata, West Bengal
  - Pfizer Investigational Site, Chennai
  - Pfizer Investigational Site, New Delhi